CLINICAL TRIAL: NCT05757180
Title: Recalling and Anticipating Specific Positive Events to Boost Resilience in Adolescents
Acronym: RASPERA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. dr. Filip Raes (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor-Investigator, Prof. dr. Filip Raes, Professor, KU Leuven
Organization: KU Leuven (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: G049019N
Record Dates: First submitted 2023-02-14; First posted 2023-03-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Specific Positive Memories; Specific Positive Future Events; Resilience; Mental Wellbeing
Keywords: adolescents; anhedonia; dampening; episodic future thinking; memory specificity; positive emotions; resilience; savoring; wellbeing
MeSH Terms: conditions — Anhedonia

STUDY DESIGN:
Intervention Model Description: A cluster randomized-controlled trial design will be used with a two (condition: PET vs. active control) x three (time-point: baseline, post-training and FU) factorial-design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Classes that will follow Positive Events Training.
  Interventions: Behavioral: Positive Events Training (PET)
- Control group (Active Comparator): Classes that will follow Bogus Control Training.
  Interventions: Behavioral: CREAtive writing Training (CREAT)

INTERVENTIONS:
Behavioral: Positive Events Training (PET) — PET is a group-based training program combining Memory Specificity Training (MEST; Raes, 2007) and Future Event Specificity Training (FEST; Dutch version of Hallford et al. (2020): Changing the Future: An initial test of Future Specificity Training). It comprises four sessions of 50 minutes each. The training is delivered in a standardized manner, using the Positive Event Training Manual developed for this study (content adapted from our MEST and FEST manuals). Following brief psychoeducation on the rationale, participants practice generating detailed specific memories and future events using neutral and positive cue-words. Participants are maximally supported and challenged by the trainer and by the other group-members to generate very specific and highly detailed memories and future events using mental imagery and drawing upon visual, olfactory, auditory and emotional elements of the events, including both contextual and sensory-perceptual details.
  Arms: Intervention group
Behavioral: CREAtive writing Training (CREAT) — CREAT follows the exact same format and length as the PET training (i.e., delivered by a trainer in group over 4 x 50-minute sessions, including homework exercises). Following brief psychoeducation on the (bogus*) rationale behind PET, participants complete a series of creative writing exercises using funny and thought-provoking writing prompts. Just as in PET, participants are maximally supported and challenged by the trainer and by the other group-members, in this case to generate completions that are as creative and funny as possible. The investigators used CREAT successfully before in an online format as a bogus control training for a memory specificity training. (*) The investigators tell participants that these creative writing exercises have been found to be beneficial for mental wellbeing, as creative writing exercises cultivate creativity and stimulate participants' imagination skills.
  Arms: Control group

SUMMARY:
Many young people are experiencing stress-related mental health problems, with some recent studies suggesting this number is increasing. Especially now, in the context of the COVID-19 pandemic, there is a significant increase in depression and anxiety in adolescents. An important way to help address this challenge is not so much to focus on trying to repair what makes young people vulnerable but to focus on building resilience. Resilience refers to the ability to successfully deal with stressful experiences. Recent research shows that being able to vividly remember and imagine positive events can buffer the negative consequences of stress, and makes a convincing case that training adolescents in recalling and anticipating positive events would promote resilience and thereby improve their mental wellbeing. And this is exactly what the current project sets out to do for the very first time. Adolescents will receive a playful group-training in school to make them better at recalling and anticipating positive events, which is expected to help them to bounce back more swiftly from challenging or otherwise stressful life events. The investigators predict that youngsters who follow our Positive Event Training will experience more positive emotions, will show improved resilience and report better mental wellbeing. The investigators will also develop a free online training protocol for teachers so that schools can provide this resilience program on their own, without the need of external professional trainers.

ELIGIBILITY:
Inclusion Criteria:

* All adolescents of the selected classes of the participating schools (12-16 years; 1st and 2nd grade of secondary school) who want to take part in the study and give informed consent (own informed consent and active parental informed consent) will be allowed to take part in the study.
* To minimize the risk of too much heterogeneity in our final sample, for instance due to context factors related to the type of education, the investigators will first recruit classes of adolescents that follow general secondary education. Future studies (after PET has been properly evaluated in this study) should also be conducted in samples of adolescents following other types of secondary education.

Exclusion Criteria:

-

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 191 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2023-05-13 (Actual); Study Completion 2023-05-13 (Actual)

PRIMARY OUTCOMES:
Change in Resilience | 1 week before the intervention, 1 week after the intervention and 2 months after the intervention.
  Connor-Davidson Resilience Scale (CD-RISC, short version) to assess resilience - This scale consists of 10 items (e.g., "Dealing with stress makes me stronger.") that are rated on a 5-point Likert scale going from 1 (not at all) to 5 (very often), with higher scores indicating higher resilience.
Change in Mental wellbeing | One week before the intervention, one week after the intervention and two months after the intervention; The SWEMWBS consists of seven statements (e.g., "I felt relaxed.") about thoughts and feelings that are scored on a 5-point Likert scale ranging from
  Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS; Stewart-Brown et al., 2009) to assess mental wellbeing - The SWEMWBS consists of seven statements (e.g., "I felt relaxed.") about thoughts and feelings that are scored on a 5-point Likert scale ranging from 1 (never) to 5 (always). Higher scores reflect higher mental wellbeing.

SECONDARY OUTCOMES:
Change in Positive affect | One week before the intervention, one week after the intervention and two months after the intervention
  Positive Affect subscale of the Positive and Negative Affect Schedule Scales (PANAS; Watson et al., 1988) to assess positive affect - The Positive Affect subscale of the PANAS consists of 10 items (words) that describe positive feelings (e.g., "excited"). Items are rated on a 5-point Likert scale going from 1 (very slightly or not at all) to 5 (extremely), where with higher scores reflecting higher positive affect.
Change in Positive affect regulation | One week before the intervention, one week after the intervention and two months after the intervention
  Dampening and Savoring subscale of the Responses to Positive Affect scale, child version (RPA-C; Bijttebier et al., 2012) to assess positive affect regulation - The RPA-C consists of items reflecting both dampening items (e.g., "When you felt happy, how often did you think: "I don't deserve this"?") and savoring items responses (e.g., "When you felt happy, how often did you notice that you felt full of energy?"). All 17 items are rated on a 4-point Likert scale ranging from 1 (not at all) to 4 (very often).
Change in Anhedonia | One week before the intervention, one week after the intervention and two months after the intervention
  Leuven Anhedonia Self-report Scale (LASS, 2nd version; Nelis, Bastin, Raes, & Bijttebier 2018) to assess symptoms of anhedonia - The 12All 12 items (e.g., "There were few things I looked forward to.") are rated on a 5-point Likert scale going from 1 (completely untrue) to 5 (completely true) with higher scores reflecting higher levels of anhedonia.
Change in Dampening | One week before the intervention, one week after the intervention and two months after the intervention
  Leuven Exeter Dampening Scale - General (LEDS, unpublished) to assess dampening.- The LEDS-G consists of 13 items (e.g., "I can only be happy if others are too.") that are rated on a 5-point Likert scale. Compared to the RPA dampening subscale, the LEDS-G aims to cover a larger variety of dampening appraisal styles.
Change in Savoring | One week before the intervention, one week after the intervention and two months after the intervention
  Savouring Items for the Four-Factor Model of the Abridged Ways Of Savoring Checklist in Response to Everyday Events (Original scale Bryant and Vernoff, 2007; Four-Factor Model Chadwick, 2012) to assess savoring. - Items (e.g., "I looked for other people to share it with.") are rated on a 7-point Likert scale going from 1 (totally disagree) to 7 (totally agree), with higher scores reflecting higher levels of savoring.
Change in Depressive symptoms and stress | One week before the intervention, one week after the intervention and two months after the intervention
  Depression, Anxiety, and Stress Scale (DASS-21; Lovibond & Lovibond, 1995) to assess basic mental health to control for baseline differences in the training groups, and to explore the generalised effect of PET on levels of depressive symptoms and stress at post-intervention and at follow-up. - The DASS-21 consists of 21 items (e.g., "I felt like my life had no meaning.") that are rated on a 4-point Likert scale going from 0 (never) to 3 (almost always).

OTHER OUTCOMES:
Change in episodic future thinking specificity (manipulation check) | One week before the intervention, one week after the intervention and two months after the intervention
  Episodic Future Thinking Test (EFT-T; Hallford et al., 2019) to assess episodic future thinking specificity. - Generated events will be coded as 0 or 1 (specific vs. non-specific) by the involved researchers.
Change in positive memory specificity (manipulation check) | One week before the intervention, one week after the intervention and two months after the intervention
  Autobiographical Memory Test (AMT, Raes et al., 2099) to assess positive memory specificity. - Generated memories will be coded as specific vs. non-specific (1 vs. 0) by the involved researchers.
Change in Pleasure | One week before the intervention, one week after the intervention and two months after the intervention
  Two single-item ratings of the anticipated/anticipatory (future) or remembered/felt pleasure (past) associated with the events participants recall/generate on the AMT and EFT-T. - 1 (not at all applicable) to 9 (strongly applicable) response rating scale presented by each generated event.
Change in Detail and mental imagery | One week before the intervention, one week after the intervention and two months after the intervention
  Two single-item ratings of level of detail and mental imagery associated with the events participants recall/generate on the AMT and EFT-T respectively. - 1 (not at all applicable) to 9 (strongly applicable) response rating scale presented by each generated event.
Change in Perceived control and likelihood | One week before the intervention, one week after the intervention and two months after the intervention
  Two single-item ratings of perceived control and perceived likelihood of occurrence associated with the events participants generate on the EFT-test (no parallel items for the AMT). - 1 (not at all applicable) to 9 (strongly applicable) response rating scale presented by each generated event.
Change in Positive feelings | One week before the intervention, one week after the intervention and two months after the intervention
  Two additional single-items ratings of anticipated/anticipatory (future) or remembered/felt positive feelings in general (past) associated with the events participants recall/generate on the AMT and EFT-T. - 1 (not at all applicable) to 9 (strongly applicable) response rating scale presented by each generated event.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Raes, Prof. dr., Principal Investigator — KU Leuven
Locations (5):
- Belgium (5):
  - Sint Lambertuscollege, Bilzen, Limburg
  - GO! Next sportschool Hasselt, Hasselt, Limburg
  - Scholen Kindsheid Jesu, Hasselt, Limburg
  - KOBOS Secundaire Scholen, Kapelle-op-den-Bos, Vlaams-Brabant
  - Pius X - instituut, Antwerp

IPD SHARING:
Plan to Share IPD: Yes
The coded, pseudonomized dataset will be uploaded in a csv format to OSF (in a restricted access repository).
Supporting Information: Study Protocol, ICF
Time Frame: The coded, pseudonomized dataset will be uploaded in a csv format to OSF (in a restricted access repository) upon publication of the research results.
Access Criteria: Coded, pseudonomized data can be shared with regulatory authorities, ethical committees, other parties that collaborate with the research team. Other researchers will only have access to the coded, pseudonomized data, and only if they agree with the confidentiality rules agreed upon within this study.

REFERENCES:
- [Background] Mojtabai R, Olfson M, Han B. National Trends in the Prevalence and Treatment of Depression in Adolescents and Young Adults. Pediatrics. 2016 Dec;138(6):e20161878. doi: 10.1542/peds.2016-1878. Epub 2016 Nov 14. PMID 27940701
- [Background] Nearchou F, Flinn C, Niland R, Subramaniam SS, Hennessy E. Exploring the Impact of COVID-19 on Mental Health Outcomes in Children and Adolescents: A Systematic Review. Int J Environ Res Public Health. 2020 Nov 16;17(22):8479. doi: 10.3390/ijerph17228479. PMID 33207689
- [Background] Jorm AF, Patten SB, Brugha TS, Mojtabai R. Has increased provision of treatment reduced the prevalence of common mental disorders? Review of the evidence from four countries. World Psychiatry. 2017 Feb;16(1):90-99. doi: 10.1002/wps.20388. PMID 28127925
- [Background] Skrove M, Romundstad P, Indredavik MS. Resilience, lifestyle and symptoms of anxiety and depression in adolescence: the Young-HUNT study. Soc Psychiatry Psychiatr Epidemiol. 2013 Mar;48(3):407-16. doi: 10.1007/s00127-012-0561-2. Epub 2012 Aug 8. PMID 22872359
- [Background] Simon-Saiz MJ, Fuentes-Chacon RM, Garrido-Abejar M, Serrano-Parra MD, Larranaga-Rubio E, Yubero-Jimenez S. Influence of resilience on health-related quality of life in adolescents. Enferm Clin (Engl Ed). 2018 Sep-Oct;28(5):283-291. doi: 10.1016/j.enfcli.2018.06.003. Epub 2018 Jul 20. English, Spanish. PMID 30037487
- [Background] Askelund AD, Schweizer S, Goodyer IM, van Harmelen AL. Positive memory specificity is associated with reduced vulnerability to depression. Nat Hum Behav. 2019 Mar;3(3):265-273. doi: 10.1038/s41562-018-0504-3. Epub 2019 Jan 14. PMID 30953005
- [Background] Speer ME, Delgado MR. Reminiscing about positive memories buffers acute stress responses. Nat Hum Behav. 2017 May;1(5):0093. doi: 10.1038/s41562-017-0093. Epub 2017 Apr 24. PMID 31482135
- [Background] Arditte Hall KA, De Raedt R, Timpano KR, Joormann J. Positive memory enhancement training for individuals with major depressive disorder. Cogn Behav Ther. 2018 Mar;47(2):155-168. doi: 10.1080/16506073.2017.1364291. Epub 2017 Aug 22. PMID 28826327
- [Background] Hallford DJ, Yeow JJE, Fountas G, Herrick CA, Raes F, D'Argembeau A. Changing the future: An initial test of Future Specificity Training (FeST). Behav Res Ther. 2020 Aug;131:103638. doi: 10.1016/j.brat.2020.103638. Epub 2020 May 7. PMID 32416495
- [Background] Tugade MM, Fredrickson BL. Resilient individuals use positive emotions to bounce back from negative emotional experiences. J Pers Soc Psychol. 2004 Feb;86(2):320-33. doi: 10.1037/0022-3514.86.2.320. PMID 14769087
- [Background] Fredrickson BL. The role of positive emotions in positive psychology. The broaden-and-build theory of positive emotions. Am Psychol. 2001 Mar;56(3):218-26. doi: 10.1037//0003-066x.56.3.218. PMID 11315248
- [Background] Nelis S, Holmes EA, Raes F. Response Styles to Positive Affect and Depression: Concurrent and Prospective Associations in a Community Sample. Cognit Ther Res. 2015;39(4):480-491. doi: 10.1007/s10608-015-9671-y. PMID 26229213
- [Background] Nelis S, Bastin M, Raes F, Bijttebier P. When Do Good Things Lift You Up? Dampening, Enhancing, and Uplifts in Relation To Depressive and Anhedonic Symptoms in Early Adolescence. J Youth Adolesc. 2018 Aug;47(8):1712-1730. doi: 10.1007/s10964-018-0880-z. Epub 2018 Jun 20. PMID 29926335
- [Background] Vinckier F, Gourion D, Mouchabac S. Anhedonia predicts poor psychosocial functioning: Results from a large cohort of patients treated for major depressive disorder by general practitioners. Eur Psychiatry. 2017 Jul;44:1-8. doi: 10.1016/j.eurpsy.2017.02.485. Epub 2017 Mar 8. PMID 28535406
- [Background] Hallford DJ, Sharma MK. Anticipatory pleasure for future experiences in schizophrenia spectrum disorders and major depression: A systematic review and meta-analysis. Br J Clin Psychol. 2019 Nov;58(4):357-383. doi: 10.1111/bjc.12218. Epub 2019 Mar 10. PMID 30854671
- [Background] Ducasse D, Loas G, Dassa D, Gramaglia C, Zeppegno P, Guillaume S, Olie E, Courtet P. Anhedonia is associated with suicidal ideation independently of depression: A meta-analysis. Depress Anxiety. 2018 May;35(5):382-392. doi: 10.1002/da.22709. Epub 2017 Dec 12. PMID 29232491
- [Background] Hallford DJ, Carmichael AM, Austin DW, Takano K, Raes F, Fuller-Tyszkiewicz M. A study protocol for a randomised trial of adjunct computerised memory specificity training (c-MeST) for major depression in youth: targeting cognitive mechanisms to enhance usual care outcomes in mental health settings. Trials. 2020 Jan 14;21(1):85. doi: 10.1186/s13063-019-4036-6. PMID 31937350
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Raes F, Williams JM, Hermans D. Reducing cognitive vulnerability to depression: a preliminary investigation of MEmory Specificity Training (MEST) in inpatients with depressive symptomatology. J Behav Ther Exp Psychiatry. 2009 Mar;40(1):24-38. doi: 10.1016/j.jbtep.2008.03.001. Epub 2008 Mar 12. PMID 18407245
- [Background] Soer R, Six Dijkstra MWMC, Bieleman HJ, Stewart RE, Reneman MF, Oosterveld FGJ, Schreurs KMG. Measurement properties and implications of the Brief Resilience Scale in healthy workers. J Occup Health. 2019 May;61(3):242-250. doi: 10.1002/1348-9585.12041. Epub 2019 Mar 22. PMID 30903648
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Stewart-Brown S, Tennant A, Tennant R, Platt S, Parkinson J, Weich S. Internal construct validity of the Warwick-Edinburgh Mental Well-being Scale (WEMWBS): a Rasch analysis using data from the Scottish Health Education Population Survey. Health Qual Life Outcomes. 2009 Feb 19;7:15. doi: 10.1186/1477-7525-7-15. PMID 19228398
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Feldman GC, Joormann J, Johnson SL. Responses to Positive Affect: A Self-Report Measure of Rumination and Dampening. Cognit Ther Res. 2008 Aug 1;32(4):507-525. doi: 10.1007/s10608-006-9083-0. PMID 20360998
- [Background] Bastin M, Nelis S, Raes F, Vasey MW, Bijttebier P. Party Pooper or Life of the Party: Dampening and Enhancing of Positive Affect in a Peer Context. J Abnorm Child Psychol. 2018 Feb;46(2):399-414. doi: 10.1007/s10802-017-0296-3. PMID 28391490
- [Background] Reijntjes A, Dekovic M, Vermande M, Telch MJ. Role of depressive symptoms in early adolescents' online emotional responding to a peer evaluation challenge. Depress Anxiety. 2009;26(2):135-46. doi: 10.1002/da.20446. PMID 19031485
- [Background] Hallford DJ, Austin DW, Takano K, Fuller-Tyszkiewicz M, Raes F. Computerized Memory Specificity Training (c-MeST) for major depression: A randomised controlled trial. Behav Res Ther. 2021 Jan;136:103783. doi: 10.1016/j.brat.2020.103783. Epub 2020 Nov 27. PMID 33291054
- [Background] Clarke A, Friede T, Putz R, Ashdown J, Martin S, Blake A, Adi Y, Parkinson J, Flynn P, Platt S, Stewart-Brown S. Warwick-Edinburgh Mental Well-being Scale (WEMWBS): validated for teenage school students in England and Scotland. A mixed methods assessment. BMC Public Health. 2011 Jun 21;11:487. doi: 10.1186/1471-2458-11-487. PMID 21693055
- [Background] Hallford DJ, Barry TJ, Austin DW, Raes F, Takano K, Klein B. Impairments in episodic future thinking for positive events and anticipatory pleasure in major depression. J Affect Disord. 2020 Jan 1;260:536-543. doi: 10.1016/j.jad.2019.09.039. Epub 2019 Sep 9. PMID 31539690
- [Background] Williams JM, Barnhofer T, Crane C, Herman D, Raes F, Watkins E, Dalgleish T. Autobiographical memory specificity and emotional disorder. Psychol Bull. 2007 Jan;133(1):122-48. doi: 10.1037/0033-2909.133.1.122. PMID 17201573
- [Background] Raes F, Hermans D, Williams JM, Demyttenaere K, Sabbe B, Pieters G, Eelen P. Reduced specificity of autobiographical memory: a mediator between rumination and ineffective social problem-solving in major depression? J Affect Disord. 2005 Aug;87(2-3):331-5. doi: 10.1016/j.jad.2005.05.004. PMID 15979154
- [Background] Bromberg U, Wiehler A, Peters J. Episodic Future Thinking Is Related to Impulsive Decision Making in Healthy Adolescents. Child Dev. 2015 Sep-Oct;86(5):1458-68. doi: 10.1111/cdev.12390. Epub 2015 Jun 25. PMID 26110500
- [Background] Bromberg U, Lobatcheva M, Peters J. Episodic future thinking reduces temporal discounting in healthy adolescents. PLoS One. 2017 Nov 22;12(11):e0188079. doi: 10.1371/journal.pone.0188079. eCollection 2017. PMID 29166658
- [Background] Sherdell L, Waugh CE, Gotlib IH. Anticipatory pleasure predicts motivation for reward in major depression. J Abnorm Psychol. 2012 Feb;121(1):51-60. doi: 10.1037/a0024945. Epub 2011 Aug 15. PMID 21842963
- [Derived] Loyen E, Bogaert L, Hallford DJ, D'Argembeau A, Raes F. Study protocol for a randomized controlled trial of the RASPERA project: recalling and anticipating specific positive events to boost resilience in adolescents. Front Public Health. 2023 Nov 24;11:1216988. doi: 10.3389/fpubh.2023.1216988. eCollection 2023. PMID 38074707